CLINICAL TRIAL: NCT07091032
Title: Building Connections Between Practices, Patients, and Community Health
Brief Title: Building Connections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Margarita Alegria, PhD, Chief, Disparities Research Unit, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2025P000661
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Cancer Colorectal; Cancer Cervix; Depression, Anxiety; Obesity
MeSH Terms: conditions — Colonic Neoplasms; Uterine Cervical Neoplasms; Depression; Anxiety Disorders; Obesity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as Usual (TAU) (Active Comparator): This comparison condition will involve treatment as usual at the clinical sites.
  Interventions: Other: Treatment as Usual
- Intervention (Experimental): The Building Connections intervention combines 3 interventions for Obesity, Cancer Screening, and Mental Health.
  Interventions: Behavioral: Building Connections Intervention

INTERVENTIONS:
Other: Treatment as Usual — This is the comparison condition, in which participants will receive treatment as usual for their conditions at the clinic.
  Arms: Treatment as Usual (TAU)
Behavioral: Building Connections Intervention — The combined Building Connections intervention incorporates three areas. Participants take part in those for which they are eligible. The obesity/weight management intervention offers coaching and support for education on evidence-based anti-obesity medications (AOM) and a lifestyle behavioral intervention offered by Community Health Workers focused on diet and physical activity. The cancer screening intervention focuses on developing workflows and systems to offer a CHW-delivered population-based intervention to improve colorectal and cervical cancer, focusing on newer screening modalities and monitoring adherence for individuals with a positive screening test result. The mental health intervention uses the evidence-based Strong Minds intervention, a 10-session psychoeducational program provided by trained community health workers with clinical supervision. The skills-based intervention uses an integrative approach aimed at improving depression, anxiety, and trauma-related symptoms.
  Arms: Intervention

SUMMARY:
Building Connections seeks to address health and healthcare inequities in socially vulnerable communities. The project will be conducted in collaboration with clinical practices across Massachusetts, serving a diverse population heavily represented in Community Clinics and Health Centers. The program will offer evidence-based interventions in obesity/weight management, cancer screening, and mental health.

ELIGIBILITY:
Inclusion Criteria:

* The general inclusion criteria involve being 18+, speaking English or Spanish, and meeting one or more of the following criteria:

Obesity: Patients with a body mass index of 30 kg/m2 or greater (i.e., obese category).

Cancer screening: Average-risk patients without recommended colorectal or cervical cancer screenings for their age group and biological sex. Specifically:

Colon Cancer (CRC) inclusion criteria: Patients aged 45-75 who are due for screenings, with last FIT longer than 1 year ago, last colonoscopy longer than 10 years ago, and last Cologuard longer than 3 years ago.

And/or

Cervical cancer inclusion criteria: Women and patients with a cervix aged 30-65 who are due for screening: with last pap longer than 3 years ago; last co-test longer than 5 years ago; last primary HPV screening longer than 5 years ago.

Mental health: Patients with moderate to severe depression or anxiety symptoms.

Exclusion Criteria:

* The general exclusion criteria are: those with current pregnancy, or the participant is cognitively impaired, not having a visit to the primary care clinic in the prior 2 years, and speaking a language other than English or Spanish.

Exclusion criteria for obesity intervention: had prior metabolic or bariatric surgery or planning to have this surgery in the next 6 months, currently enrolled in an intensive lifestyle program.

Exclusion criteria for cancer screening intervention include:

Colon Cancer (CRC) exclusion criteria: has colorectal cancer documented in the problem list; has ulcerative colitis or Crohn's disease documented in the problem list

Cervical cancer exclusion criteria: has cervical cancer documented in the problem list; has had a prior hysterectomy.

Exclusion criteria for mental health: include patients with active suicidality, active substance use disorder, a history of schizophrenia or bipolar disorder, or who are already receiving behavioral health care (therapy sessions in the past 3 months or an appointment upcoming in the next month).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3600 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Self-reported height/weight for Body Mass Index (BMI) | Baseline, month 6, and month 12
  Calculation of Body Mass Index
Rate of cancer screening test completion | Baseline, month 6, month 12
  Number of eligible people who complete a screening test out of total eligible
Computerized Adaptive Testing (CAT) of Mental Health (MH) | Baseline, month 6, month 12
  CAT-MH Depression/MDD and Anxiety

SECONDARY OUTCOMES:
Rapid Prime Diet Quality Score Screener (rPDQS) | Baseline, month 6, month 12
  The Rapid Prime Diet Quality Score Screener (rPDQS) is a 13-item measure about past month consumption of food, categorized by type (less than once per week to twice per day or more). A logic system assigns points to each item (0 'unhealthy dietary pattern' to 2 'healthy dietary pattern'). Total scores are calculated as the sum of all items (range 0 to 26), and higher scores represent healthier dietary patterns.
Cancer screening test type | Baseline, month 6, month 12
  Screening test type used by people who completed a screening
World Health Organization Disability Assessment Schedule (WHODAS) 2.0 | Baseline, month 6, month 12
  The World Health Organization Disability Assessment Schedule (WHODAS) 2.0 is a 12-item measure of difficulties performing activities in six domains of daily life (1 'None' to 5 'Extreme or cannot do'). Total scores are calculated as the sum of all items (range 12 to 60) and higher scores indicate higher disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Disparities Research Unit, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No